CLINICAL TRIAL: NCT06185712
Title: The Impact of Nurse-led Disease Management Education on Outcomes of Patients With Ankylosing Spondylitis: Randomised Controlled Trial
Brief Title: Patient Education in Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeliha Tülek (Other)
Responsible Party: Sponsor-Investigator, Zeliha Tülek, RN, Prof, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Disease management in AS
Record Dates: First submitted 2023-12-07; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Ankylosing Spondylitis
Keywords: Patient Education; Nursing; Rheumatology
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led disease management education (Experimental): Individual patient education was provided, and patients were followed up by telephone at two-week intervals beginning the week after their clinic visit.
  Interventions: Behavioral: Nurse-led disease management education
- Control Group (No Intervention): No interventions were performed other than routine clinical procedures.

INTERVENTIONS:
Behavioral: Nurse-led disease management education — Nurse-led disease management education was applied to the intervention group
  Arms: Nurse-led disease management education

SUMMARY:
This study was carried out to investigate the effect of a nurse-led disease management education program in AS on patient compliance, disease activity, functional capacity, kinesiophobia, and quality of life. A total of 122 patients diagnosed with AS according to the modified New York criteria were included in the study. The intervention group received nurse-led individualized disease management education. In the control group, no interventions were performed other than routine clinical procedures.

DETAILED DESCRIPTION:
This study was carried out to investigate the effect of a nurse-led disease management education program in AS on patient compliance, disease activity, functional capacity, kinesiophobia, and quality of life. A total of 122 patients diagnosed with AS according to the modified New York criteria were included in the study. The intervention group received nurse-led individualized disease management education. After the education, the group was contacted by telephone six times for 12 weeks to monitor the results. Patient education was provided through booklets and videos. In the control group, no interventions were performed other than routine clinical procedures.Patients were assessed using the same scales at baseline and end of the week 12.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years
* Have a clinical diagnosis AS according to the modified New York criteria
* Receiving TNF-α inhibitor treatment.

Exclusion Criteria:

* Communication difficulties
* Illiterates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in scores Bath Ankylosing Spondylitis Disease Activity Index | 12 weeks
  Disease Activity will be evaluated by Bath Ankylosing Spondylitis Disease Activity Index. There are 6 questions in the scale that examine the symptoms of joint pain, fatigue and morning stiffness. Using a visual analog scale, patients are asked to give points (0-10 points) for each question according to the severity of the symptoms (0 = no symptoms, 10 = very severe). The scale score is calculated by taking the average score of the last two questions regarding morning stiffness, adding the scores from the first four questions, and dividing the result by 5. An increase in the scale score is considered as an increase in disease activity, and a decrease in the score is considered as a decrease in disease activity.
Change in scores Bath Ankylosing Spondylitis Functional Index | 12 weeks
  Functional Status will be evaluated by Bath Ankylosing Spondylitis Functional Index. Patients are asked to rate how difficult they are doing each activity on a scale of 0-10 (0 = easy, 10 = impossible). Scale scoring is calculated by adding the scores of all questions and dividing by 10. An increase in the BASFI score is considered as a decrease in functional capacity.
Change in scores Compliance Questionnaire on Rheumatology | 12 weeks
  Treatment compliance will be evaluated by Compliance Questionnaire on Rheumatology.It consists of 19 items. The scores obtained from the scale vary between 0-100 points, and higher scores indicate increased compliance, while lower scores indicate decreased compliance.
Change in scores Ankylosing Spondylitis Quality of Life Scale | 12 weeks
  Quality of life will be evaluated by Ankylosing Spondylitis Quality of Life Scale. In the scale where disease symptoms, functional status and concerns about the disease are questioned, one of the options "Yes" or "No" is selected for each question (Yes = 1, No = 0), and the scale score varies between 0-18 points. An increase in the score is considered as a decrease in the quality of life.
Change in scores Tampa Scale for Kinesiophobia | 12 weeks
  Kinesiophobia will be evaluated by Tampa Scale for Kinesiophobia. The scale score is calculated by summing the scores from each question and varies between 17-68 points. An increase in the scale score is considered as an increase in the fear of movement / injury.

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Dağ, RN, PhD, Principal Investigator — Istanbul University - Cerrhapasa; Zeliha Tulek, RN, Prof, Study Director — Istanbul University - Cerrhapasa; Emire Seyahi, MD, Prof, Study Chair — Istanbul University - Cerrhapasa
Locations (1):
- Istanbul University-Cerrahpasa Cerrahpasa Medical Faculty Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duruoz MT, Doward L, Turan Y, Cerrahoglu L, Yurtkuran M, Calis M, Tas N, Ozgocmen S, Yoleri O, Durmaz B, Oncel S, Tuncer T, Sendur O, Birtane M, Tuzun F, Bingol U, Kirnap M, Celik Erturk G, Ardicoglu O, Memis A, Atamaz F, Kizil R, Kacar C, Gurer G, Uzunca K, Sari H. Translation and validation of the Turkish version of the Ankylosing Spondylitis Quality of Life (ASQOL) questionnaire. Rheumatol Int. 2013 Nov;33(11):2717-22. doi: 10.1007/s00296-013-2796-y. Epub 2013 Jun 14. PMID 23765201
- [Background] Garrett S, Jenkinson T, Kennedy LG, Whitelock H, Gaisford P, Calin A. A new approach to defining disease status in ankylosing spondylitis: the Bath Ankylosing Spondylitis Disease Activity Index. J Rheumatol. 1994 Dec;21(12):2286-91. PMID 7699630